CLINICAL TRIAL: NCT03411031
Title: A Randomized Parallel Phase 2 Study of Elotuzumab Plus Lenalidomide (Elo/Rev) for the Treatment of Serologic Relapse/Progression While on Lenalidomide Maintenance for Multiple Myeloma
Brief Title: Elotuzumab Plus Lenalidomide (Elo/Rev) for Serologic Relapse/Progression While on Lenalidomide
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor no longer providing drug
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19197; NCI-2018-00891 (Other: NCI)
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
Keywords: lenalidomide maintenance; hematopoietic cell transplantation; serologic relapse
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A: Elotuzumab + Lenalidomide at 25 mg (Active Comparator): Elotuzumab 10 mg/kg intravenously (IV) weekly (days 1, 8, 15 and 22) for 2 cycles, then 20 mg/kg every 4 weeks. Dexamethasone will be administered as premedication for elotuzumab.
  Lenalidomide 25 mg by mouth (PO) daily days 1-21 out of a 28-day schedule.
  Interventions: Drug: Elotuzumab; Drug: Lenalidomide; Drug: Dexamethasone
- B: Elotuzumab + Lenalidomide at 10 mg (Active Comparator): Elotuzumab 10 mg/kg IV weekly (days 1, 8, 15 and 22) for 2 cycles, then 20 mg/kg every 4 weeks. Dexamethasone will be administered as premedication for elotuzumab.
  Lenalidomide 10 mg PO daily days 1-21 out of a 28-day schedule.
  Interventions: Drug: Elotuzumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elotuzumab — Elotuzumab according to dosing schedule outlined in treatment arms.
  Other Names: Empliciti™; BMS-901608; HuLuc63
Drug: Lenalidomide — Lenalidomide according to dosing schedule outlined in treatment arms.
  Other Names: REVLIMID®; thalidomide analogue
Drug: Dexamethasone — Dexamethasone is a commercially available drug. The description, how supplied, and storage instructions for dexamethasone product are found in the prescribing information.
  During the study, dexamethasone will be administered as premedication for elotuzumab as indicated in the package insert.
  Other Names: Decadron

SUMMARY:
The purpose of this study is determine Time-to-Progression with elotuzumab plus lenalidomide when elotuzumab is added to multiple myeloma participants with serologic relapse/progression while receiving lenalidomide maintenance for each study arm.

DETAILED DESCRIPTION:
This is a randomized parallel 2-cohort phase 2 study of elotuzumab given at 10 mg/kg weekly during induction in combination with lenalidomide (either 25 mg or 10 mg) in patients with multiple myeloma who progress or relapse serologically while on single agent lenalidomide maintenance.

The combination therapy with elotuzumab and lenalidomide will be continued until further progression of myeloma (based on response criteria) or intolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who demonstrate evidence of serologic relapse/progression while on lenalidomide maintenance given as part of first line therapy (including upfront high-dose chemotherapy followed by autologous hematopoietic cell transplantation (HCT)) without symptomatic relapse/progression. Lenalidomide maintenance is defined as single agent lenalidomide therapy of any doses up to 10 mg PO daily for up to 28 days (28-day cycle).
* Male or female patients aged ≥ 18 years old
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Measurable disease as outlined in protocol guidelines
* Participants must meet laboratory criteria as outlined in protocol guidelines

Exclusion Criteria:

* Prior Elotuzumab
* Patients with clinical relapse/progression as per the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma defined as one or more of the following criteria:

  * Development of new soft tissue plasmacytomas or bone lesions (osteoporotic fractures do not constitute progression)
  * Definite increase in the size of existing plasmacytomas or bone lesions. A definite increase is defined as a 50% (and ≥1 cm) increase as measured serially of the measurable lesion
  * Hypercalcemia (>11 mg/dL);
  * Decrease in hemoglobin of ≥2 g/dL not related to therapy or other non-myeloma-related conditions;
  * Rise in serum creatinine by 2 mg/dL or more from the start of the therapy and attributable to myeloma
  * Hyperviscosity related to serum paraprotein
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy testing within 7 days prior to the administration of drug.
* Male patients whose sexual partners are WOCBP not using effective birth control
* Patients with a prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Patients with known positivity for human immunodeficiency virus (HIV)) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with a diagnosis of POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or plasma cell leukemia (> 2.0 × 10^9/L circulating plasma cells by standard differential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Elotuzumab + Lenalidomide at 25 mg: Elotuzumab 10 mg/kg intravenously (IV) weekly (days 1, 8, 15 and 22) for 2 cycles, then 20 mg/kg every 4 weeks. Dexamethasone will be administered as premedication for elotuzumab.
  Lenalidomide 25 mg by mouth (PO) daily days 1-21 out of a 28-day schedule.
  Elotuzumab: Elotuzumab according to dosing schedule outlined in treatment arms.
  Lenalidomide: Lenalidomide according to dosing schedule outlined in treatment arms.
  Dexamethasone: Dexamethasone is a commercially available drug. The description, how supplied, and storage instructions for dexamethasone product are found in the prescribing information.
  During the study, dexamethasone will be administered as premedication for elotuzumab as indicated in the package insert.
- B: Elotuzumab + Lenalidomide at 10 mg: Elotuzumab 10 mg/kg IV weekly (days 1, 8, 15 and 22) for 2 cycles, then 20 mg/kg every 4 weeks. Dexamethasone will be administered as premedication for elotuzumab.
  Lenalidomide 10 mg PO daily days 1-21 out of a 28-day schedule.
  Elotuzumab: Elotuzumab according to dosing schedule outlined in treatment arms.
  Lenalidomide: Lenalidomide according to dosing schedule outlined in treatment arms.
  Dexamethasone: Dexamethasone is a commercially available drug. The description, how supplied, and storage instructions for dexamethasone product are found in the prescribing information.
  During the study, dexamethasone will be administered as premedication for elotuzumab as indicated in the package insert.
Period: Overall Study
Arm/Group | A: Elotuzumab + Lenalidomide at 25 mg | B: Elotuzumab + Lenalidomide at 10 mg
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Elotuzumab + Lenalidomide at 25 mg | B: Elotuzumab + Lenalidomide at 10 mg | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time of randomization to date of death from any cause, date of relapse/progression, or the last follow-up date, whichever comes first. The Kaplan-Meier method will be used to estimate PFS for each Study Arm. The method of Brookmeyer and Crowley will be used to construct 95% confidence interval.
Time Frame: An average of 8 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Elotuzumab + Lenalidomide at 25 mg | B: Elotuzumab + Lenalidomide at 10 mg
Number analyzed (Participants) | 9 | 9
percentage of participants | 11.1 [0.1 to 38.8] | 22.2 [3.4 to 51.3]

2. Secondary Outcome: Overall Response
Description: Overall response with elotuzumab and lenalidomide for each study arm. Overall Response is defined as best Overall Response, as Complete Response or Partial Response. Response will be assessed per the uniform response criteria of the International Myeloma Working Group(IMWG). Myeloma participants enrolled in this clinical study will be assessed for disease response after every cycle. Complete Response= Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates; Partial Response= ≥50% reduction of serum M-protein plus reduction in 24 h urinary M-protein by ≥90% or to <200 mg per 24 h;
Time Frame: Up to 60 days post last study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | A: Elotuzumab + Lenalidomide at 25 mg | B: Elotuzumab + Lenalidomide at 10 mg
Number analyzed (Participants) | 9 | 9
Participants | 1 | 2

3. Secondary Outcome: Minimum Response (MR)
Description: Minimum response (MR) or better with elotuzumab and lenalidomide for each study arm. The Consensus on Uniform Reporting of Response will be used to evaluate response. Myeloma participants enrolled in this clinical study will be assessed for disease response after every cycle.
Time Frame: Up to 60 days post last study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | A: Elotuzumab + Lenalidomide at 25 mg | B: Elotuzumab + Lenalidomide at 10 mg
Number analyzed (Participants) | 9 | 9
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from cycle 1, day 1, and only while the participants were on study treatment only for up to a total of 12 months.
Arm/Group | A: Elotuzumab + Lenalidomide at 25 mg | B: Elotuzumab + Lenalidomide at 10 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9 | 0/9
Other Adverse Events (participants affected / at risk) | 2/9 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Elotuzumab + Lenalidomide at 25 mg (N=9) | B: Elotuzumab + Lenalidomide at 10 mg (N=9)
Fever (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Lung Infection - Probable Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Elotuzumab + Lenalidomide at 25 mg (N=9) | B: Elotuzumab + Lenalidomide at 10 mg (N=9)
Fatigue (General disorders) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT03411031/Prot_SAP_000.pdf